CLINICAL TRIAL: NCT04335214
Title: Advance Care Planning Among Older People From Moroccon Origin in Belgium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B670201942542
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-05

CONDITIONS: Advance Care Planning; Ethnic Minorities; Moroccans; Advance Medical Directives; Muslims; Living Will

STUDY DESIGN:
Intervention Model Description: one to one interviews
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interview (Other): One to one interview with older people from moroccon origin in Belgium
  Interventions: Other: one to one interview

INTERVENTIONS:
Other: one to one interview — one to one interviews with older people from moroccon origin in Belgium

SUMMARY:
Advance care planning (ACP) enables individuals to define goals and preferences for future medical treatment and care, to discuss these goals and preferences with family and health-care providers, and to record and review these preferences if appropriate. Research has shown that most Western patients express the need about what ACP entails. Ethnicity creates an important cultural impact on how people look at life and death, so that there is an influence on making decisions about end-of-life care.

The moroccan ethnic group is one of the largest visible non-Western minority groups in Western countries. Studies on how ACP is perceived among patients from moroccon origin are lacking. The objective of this study is exploring the knowledge, experiences, point of views, preferences, attitudes, facilitators and barriers concerning advance care planning of older people from moroccan origin in Belgium. Semi-structured interviews (in the native moroccan/arabic language) will be used.

ELIGIBILITY:
Inclusion Criteria:

* People with Moroccan origin who live in Belgium and are older than 65 years and who have also given informed consent to participate in this qualitative interview study

Exclusion Criteria:

* Patients who are terminal ill which means having a life-limiting disease with irreversible decline and who are actively dying (actively dying is related to patients with days of survival). (41)
* people who have cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Knowledge, experiences, views, preferences, barriers and facilitators about advance care planning from older people from moroccon origin in Belgium | 18 months
  This is a qualitative study. We've developed a semi-structured interview guide with the folowing questions: What do you know in relation to advance care planning? Have you yourself ever thought or looked up about your future healthcare? What do you think about advance care planning now for future? What are the advantages and disadvantages? In your opinion, what makes it easier or harder to talk about advance care planning?

CONTACTS AND LOCATIONS:
Overall Officials: Hakki Demirkapu, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Faculteit Geneeskunde en Farmacie, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
data will be with the prinicipal investigator

REFERENCES:
- [Derived] Demirkapu H, Hajji R, Chater B, De Maesschalck S, Van den Block L, De Vleminck A, Devroey D. Advance care planning among older adults of Moroccan origin: An interview-based study. Patient Educ Couns. 2023 Aug;113:107794. doi: 10.1016/j.pec.2023.107794. Epub 2023 May 13. PMID 37196404